CLINICAL TRIAL: NCT04183517
Title: A Two-part Pharmacokinetic Study of PXS-5382A in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PXS-5382A-102
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasted (Experimental): PXS-5382A administered as a single dose in the fasted state
  Interventions: Drug: PXS-5382A
- Fed (Experimental): PXS-5382A administered as a single dose in the fed state
  Interventions: Drug: PXS-5382A
- Twice daily (Experimental): PXS-5382A administered twice daily for 5 days in the fed state
  Interventions: Drug: PXS-5382A

INTERVENTIONS:
Drug: PXS-5382A — Orally once daily or twice daily

SUMMARY:
This is a Phase I, open-label, two-part in healthy adult males. There will be up to 12 subjects with 6 subjects in each part of the study. Subjects from Part A are eligible to participate in Part B.

For Part A, each of the 6 subjects will complete two periods of the study with washout period of 7 days between. Each subject during participation in the study will receive a dose of PXS 5382A orally in a fed state and a fasted state.

For Part B, repeated oral BID administration of PXS-5382A will be performed in the Fed state and dose will be dependent on analysis of Part A.

In both part A and B PK, PD and safety assessments will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, aged between 18 and 60 years (inclusive).
2. Eligibility of the subjects based on clinical history, physical examination, ECG and Lab results
3. BMI between 18.5 kg/m2 and 30.0 kg/m2 inclusive.
4. No clinically relevant abnormality in an ECG; QTcF (Fridericia's corrected QT) ≤ 450 ms, PR interval of 120-210 ms and a QRS duration ≤ 120 ms.
5. Adequate venous access in the left or right arm to allow dosing and collection of a number of blood samples.
6. Male subjects with female partners of childbearing potential may be enrolled if they:

   1. are documented to be surgically sterile (vasectomy at least six months prior to dosing), or
   2. practice true abstinence for 30 days after the study drug administration, or
   3. agree to use a barrier method of contraception (e.g. condom) from Screening and until 30 days after administration of the study. Additionally, the female partner must use a highly effective hormonal method, such as birth control pills, patches, implants or injections; or used an intra uterine device (IUD).
   4. Contraceptive requirements do not apply to subjects who are exclusively in same-sex relationships.
7. Have given written informed consent to participate in this study in accordance with local regulations.

Exclusion Criteria:

1. Clinically significant abnormal findings on the physical examination, medical history, ECG or laboratory results as deemed by the PI (or delegate).
2. Clinically significant gastrointestinal, renal, hepatic, neurologic, haematologic (including thalassaemia), endocrine, oncologic, pulmonary, immunologic, psychiatric, skin or cardiovascular disease or any other condition, which, in the opinion of the PI (or delegate), would jeopardise the safety of the subject or impacted the validity of the study results.
3. History of significant drug allergies or significant allergic reaction or suffer from clinically significant systemic allergic disease. Mild hay fever is acceptable.
4. Evidence of abnormal wound healing (e.g. hypertrophic scars) as the result of surgery or trauma as deemed by the PI or delegate.
5. Have received or are anticipated to receive any prescription systemic or topical medication, or any over the counter, supplements, complementary or alternative medicine 7 days prior to the start of dosing or within 5 half-lives of the drug whichever is longer (excluding paracetamol).
6. Systolic BP < 90 or > 140 mmHg, diastolic BP < 40 or > 90 mmHg and HR < 40 or > 100 beats per minute (BPM).
7. ALT, AST or total bilirubin > 1.5x ULN.
8. Gilbert's syndrome sufferers are not eligible.
9. Evidence of significant renal insufficiency, as indicated by an estimated creatinine clearance using the Cockcroft-Gault formula of less than 80 mL/min at Screening.
10. Positive Screening test for Hepatitis B surface antigen or Hepatitis C antibody or human immunodeficiency virus (HIV)
11. Any condition directly or indirectly caused by or associated with Transmissible Spongiform Encephalopathy (TSE) Creutzfeldt-Jakob Disease (CJD) variant Creutzfeldt-Jakob Disease (vCJD) or new variant Creutzfeldt-Jakob Disease (nvCJD)
12. History of drug abuse in the last 2 years.
13. Males who regularly drink more than four (4) units of alcohol daily (1 unit = 285 mL beer (4.9% Alc./Vol), 100 mL wine (12% Alc./Vol), 30 mL spirit (40% Alc./Vol)).
14. Use nicotine-containing products (e.g., cigarettes, e-cigarettes, cigars, chewing tobacco, snuff) within 6 weeks before screening and were unable to abstain from using these products until study completion.
15. Unable to abstain from consuming caffeine and/or xanthine products (i.e., coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.) for defined periods (eg, to the clinical facility).
16. Consumption of:

    1. Grapefruit, grapefruit juice, star fruit, oranges, orange juice, Seville oranges (CYP450 enzymes) within 7 days prior to administration of the study drug up to Exit Evaluation visit.
    2. Poppy seeds and poppy seed products within 7 days prior to administration of the study drug up to Exit Evaluation visit.
    3. Alcohol within 48 hours prior to administration of study drug up to Exit Evaluation visit.
17. Positive urine screen for drugs of abuse and alcohol breath test at screening and study check-in. Subjects may undergo a repeat urine drug screen or alcohol breath test at the discretion of the PI (or delegate).
18. Receipt of blood or blood products, or loss or donation of 450 mL or more of blood within 90 days before the first dose administration.
19. Have dietary restrictions that preclude the consumption of the required high-fat meal in Part A.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Cmax after oral administration of PXS-5382A | 6 days
  Maximum plasma concentration
Tmax after oral administration of PXS-5382A | 6 days
  Time of the observed maximum plasma concentration
AUC0-inf of PXS-5382A | 6 days
  Area under the plasma concentration-time curve (AUC) from time zero extrapolated to infinity
t1/2 of PXS-5382A | 6 days
  Terminal plasma elimination half-life

SECONDARY OUTCOMES:
Maximum percentage inhibition plasma LOXL2 of PXS-5382A | 6 days
  Maximum measured plasma LOXL2 target engagement following PXS-5382A administration
Incidence and severity of Adverse Events | 6 days
  A treatment-emergent adverse events (TEAE) will be summarized by treatment and overall, and summarized for each treatment by severity and relationship to study drug. All TEAEs leading to withdrawal, or SAEs, will be summarized.
Number of subjects with clinical laboratory test abnormalities | 6 days
  The clinical laboratory will include hematology (hematocrit, hemoglobin, mean cell hemoglobin, mean cell hemoglobin concentration, mean cell volume, platelet count, red blood cell count, white blood cell count), clinical chemistry (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, blood urea nitrogen, calcium, chloride, cholesterol, creatinine, creatine phosphokinase, direct bilirubin, estimated glomerular filtration rate, gamma glutamyl transferase, glucose. inorganic phosphate, iron, lactate dehydrogenase, phosphorus, potassium, sodium, total bilirubin, total CO2, total protein, triglyceride, urea, uric acid), and urinalysis (bilirubin, blood, color and appearance, glucose, ketones, leukocyte esterase, nitrite, pH, protein, specific gravity, urobilinogen, microscopic examination, electrolytes). Abnormality will be determined by the investigator.
Number of subjects with vital signs abnormalities | 6 days
  The vital sign will include blood pressure (mmHg), pulse rate (bpm), respiratory rate (breaths/min), and body temperature (degree Celsius). Abnormality will be determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Molga, MBBS, Principal Investigator — CMAX Ltd
Locations (1):
- CMAX, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No